CLINICAL TRIAL: NCT03148327
Title: Randomized Phase I/II Study of Ablative Radiotherapy +/- MEDI 4736 (Durvalumab) for Medically Inoperable Early-Stage Non-Small Cell Lung Cancer
Brief Title: Astra Zeneca (Immuno Stereotactic Ablative Body Radiotherapy) ISABR Study: Randomized Phase I/II Study of Stereotactic Body Radiotherapy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-000004; NCI-2017-00954 (Registry Identifier: CTRP)
Record Dates: First submitted 2017-05-03; First posted 2017-05-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Regimen A: Phase I (Experimental): The intervention will be looking at radiotherapy + drug Durvalumab (MEDI 4736)
  Interventions: Drug: Durvalumab (MEDI 4736); Radiation: Radiotherapy
- Regimen A: Phase II (Experimental): The intervention will be looking at radiotherapy + drug Durvalumab (MEDI 4736)
  Interventions: Drug: Durvalumab (MEDI 4736); Radiation: Radiotherapy
- Regimen B: Phase II (Active Comparator): Radiotherapy alone
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: Durvalumab (MEDI 4736) — Early studies has shown to possibly reduce the growth of certain types of lung cancer
  Arms: Regimen A: Phase I; Regimen A: Phase II
Radiation: Radiotherapy — Stereotactic Body Radiation Therapy (SABR)

SUMMARY:
This study uses durvalumab (MEDI 4736), an experimental type of drug made by Astra Zeneca Pharmaceuticals, (limited partnership) LP, which in early studies has shown to possibly reduce the growth of certain types of lung cancer. The Investigators will enroll up to 105 subjects into the study. After an initial safety sample of 15 individuals receiving durvalumab (MEDI 4736) and Stereotactic Ablative Body Radiotherapy (SABR), if it is shown to be safe to administer this combination of therapies, the next enrolled subjects will be randomized in a 1:1 fashion (each subject with a "50-50 chance" like the flip of a coin) to receive either SABR and durvalumab (MEDI 4736), or SABR alone.

Once treatment is completed, all subjects will return to the University of California at Los Angeles (UCLA) for regular follow-up visits to check on their health and outcomes. At visits both prior to and after treatment special blood samples will be drawn to be studied by UCLA scientists to look into the basic science aspects of how durvalumab (MEDI 4736) and radiation work in the body. It is hoped that we will learn more about the basic safety and science of durvalumab (MEDI 4736) combined with Stereotactic Ablative Body Radiotherapy (SABR) vs. SABR alone, while extending the life and quality of life of these subjects.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized phase II study with a phase I safety lead in. Patients in this study will undergo radiation therapy alone or in combination with durvalumab (MEDI 4736). Patients eligible for treatment must be diagnosed with node negative, non-metastatic, biopsy- proven early-stage NSCLC and be ineligible for surgical resection or refuse surgical resection.

Enrollment will begin with a phase I lead in evaluating radiation therapy with durvalumab (MEDI 4736). (Regimen A) to ensure general safety of this combination and specifically relating to pulmonary toxicity (pneumonitis), cardiac toxicity (pericarditis) and gastrointestinal toxicity (esophagitis, gastritis, enterocolitis). Following initial demonstration of safety, enrollment to the phase II component with 1:1 randomization to radiation therapy and durvalumab (MEDI 4736), (Regimen A) or radiation therapy alone (Regimen B) will be performed with stratification only based on T-stage (Tumor) (T1 versus T2). A total of 90 patients will be randomized in the phase II component.

Regimen A:

Durvalumab (MEDI 4736), at 1500 mg via IV infusion will be delivered on day -5 of therapy. Radiation therapy will start on Day 0 ±5 from the first infusion of durvalumab (MEDI 4736) and patients will receive 3, 4, or 10 fractions of radiation therapy to a total dose of 54 Grays (Gy), 50Gy, or 65Gy, respectively.

Starting on day 23 (28 days post first durvalumab (MEDI 4736), infusion), durvalumab (MEDI 4736), 1500mg IV q4weeks will be delivered for up to 4 additional cycles or until progression, toxicity or withdrawal from study.

Regimen B:

Patients will receive radiation therapy alone of 3, 4, or 10 fractions to a total dose of 54Gy, 50Gy, or 65Gy, respectively. Regimen B patients will not receive durvalumab (MEDI 4736) and will only receive radiation therapy.

Safety review will continue to occur on an ongoing basis. Should the rates of grade 3 treatment-related pulmonary toxicity (defined as pneumonitis), cardiac toxicity (defined as pericarditis) or gastrointestinal toxicity (defined as esophagitis, gastritis or enter colitis) be observed at a frequency greater than 15%, accrual will be halted and study will be re-evaluated. Should any patient have ≥ grade 4 treatment-related adverse effects, accrual will be halted and study will be re-evaluated Follow-up Routine surveillance computerized axial tomography (CT) imaging of the chest, abdomen, and pelvis will be performed starting at 12 weeks after completion of radiation in both treatment groups to allow for primary endpoint assessment. Routine CT imaging surveillance will continue per standard of care. Patients will also be followed clinically with history and physical examinations, vitals signs, and laboratory examinations as indicated.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects must fulfill all of the following criteria:

1. Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluation.
2. Newly diagnosed, untreated, biopsy proven non-small cell lung cancer.
3. Medically inoperable or patient refusal to surgery as defined by any single of the following criteria: a. Determined unfit for surgery by thoracic surgeon or radiation oncologist as documented in the medical record b. Pulmonary function test (PFTS) showing Forced Expiratory Volume in the first second (FEV1) ≤ 1.2 L or diffusing Lung Capacity (DLC) <60%, c. Poor exercise tolerance or failed pre-operative cardiac work-up, d. Patient refusal to undergo definitive surgery as documented in clinical note by a surgeon, pulmonologist, medical oncologist, or radiation oncologist.
4. Clinically stage I disease by American Joint Committee on Cancer (AJCC) 7th edition. (N0, M0, T stages T1-T2a) or patients with stage T2bN0M0 (clinical stage IIA) disease who are medically unfit for standard of care chemotherapy as documented by a medical oncologist or radiation oncologist, or who refuse standard of care chemotherapy as documented by a medical oncologist or radiation oncologist.
5. Age > 18 years at time of study entry.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
7. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥ 9.0 g/dL.
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3).
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3).
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). <<This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
   * aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/ alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN.
   * Serum creatinine creatinine clearance (CL) >40 mL/min by the Cockcroft-Gault formula (Cockcroft and

   Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min)

   = Weight (kg) x (140 - Age) . 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min)

   = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
8. Female subjects must either be of non-reproductive potential (i.e. post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
9. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. ECOG Performance status >1.
2. Patients with metastatic or node positive NSCLC.
3. Patients with prior radiation therapy to the same bronchopulmonary segment.
4. History of automimmune disease including myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematous, rheumatoid arthritis, inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), vascular thrombosis associated with antiphospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, or glomerulonephritis.

   a. However, patients with type 1 diabetes mellitus, vitiligo, alopecia, hypothyroidism requiring hormone replacement, Graves disease, or skin disorders not requiring systemic treatment are permitted to enroll.
5. Patients with history of idiopathic pulmonary fibrosis, idiopathic pneumonitis, drug induced pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
6. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
7. Participation in another clinical study with an investigational product during the last 6 months.
8. Any previous treatment with a Programmed Death-1 (PD1) or Programmed Death-Ligand 1(PD-L1) inhibitor, including durvalumab, and therapeutic anticancer vaccine.
9. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ.
10. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.
11. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
12. Any unresolved ≥ Grade 2 pulmonary toxicity from previous anti-cancer therapy.
13. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
14. History of primary immunodeficiency.
15. History of allogeneic organ transplant.
16. History of hypersensitivity to durvalumab or any excipient.
17. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
18. Known history of previous clinical diagnosis of tuberculosis.
19. History of leptomeningeal carcinomatosis.
20. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
21. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
22. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
23. Subjects with uncontrolled seizures. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: The number and severity of study participants' treatment-related adverse events as assessed by CTCAE v4.0. | 4 months
  the safety and tolerability associated with radiation therapy and durvalumab (MEDI 4736)
Phase II: Median Progression-Free Survival | 2 year
  Progression Free Survival for patients treated with radiation therapy with and without durvalumab (MEDI 4736) will be determined by both the 2-year progression free survival rate (percentage) and the median progression free survival (in years).

SECONDARY OUTCOMES:
Overall survival | 2 year
  the efficacy of radiation therapy and durvalumab in terms of overall survival
Primary Tumor Control | 2 year
  the efficacy of radiation therapy and durvalumab in terms of primary tumor control
Intralobar recurrence rates | 2 year
  the efficacy of radiation therapy and durvalumab in terms of intralobar recurrence rates
mediastinal recurrences | 2 year
  the efficacy of radiation therapy and durvalumab in terms of mediastinal recurrences
hilar and mediastinal recurrences | 2 year
  the efficacy of radiation therapy and durvalumab in terms of hilar and mediastinal recurrences
rate of distant recurrences | 2 years
  the efficacy of radiation therapy and durvalumab (MEDI 4736) in terms of the rate of distant recurrences
rates of grade 3 or higher non-hematological toxicities | 2 years
  rates of grade 3 or higher non-hematological toxicities with the combination of radiation therapy and durvalumab MEDI 4736)

OTHER OUTCOMES:
germline mutations as indicators | 2 years
  Germline mutations as determined by DNA sequencing will be studied to see if these mutations can predict a patients' response to treatment and treatment-related toxicities.
nonsynonymous mutational load and intratumoral heterogeneity as indicators | 2 years
  Tumor genetics (nonsynomonous mutational load and intratumoral heterogeneity) will be evaluated as possible indicators for clinical outcome (progression-free survival, overall survival, and toxicity) in patients receiving radiation therapy alone and patients treated with radiation therapy with durvalumab (MEDI 4736) .
Changes to circulating lymphocytes as indicators | 2 years
  changes to circulating lymphocytes including cluster of differentiation 8 (CD-8), Tumor (T)-regulatory cells, and myeloid suppressor cells before, during and after radiation therapy alone or in combination with durvalumab (MEDI 4736) and correlations with progression free-survival, overall survival and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ann Raldow, MD, Principal Investigator — Associate Professor
Locations (4):
- United States (3):
  - Jonsson Comprehensieve Cancer Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
- Peter MacCallum Cancer Centre, Melbourne E., Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu TC, Stube A, Felix C, Oseguera D, Romero T, Goldman J, Garon EB, Lee JM, Glaspy J, Lisberg AE, Rusthoven CG, Camidge DR, Siva S, Solomon B, Lee A, Tenn SE, Shaverdian N, Steinberg ML, Raldow AC, Lee P. Safety and Efficacy Results From iSABR, a Phase 1 Study of Stereotactic ABlative Radiotherapy in Combination With Durvalumab for Early-Stage Medically Inoperable Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2023 Sep 1;117(1):118-122. doi: 10.1016/j.ijrobp.2023.03.069. Epub 2023 Apr 5. No abstract available. PMID 37023987